CLINICAL TRIAL: NCT06650709
Title: A Phase 2, Proof of Concept Trial Investigating the Safety and Efficacy of the Neoadjuvant Triplet Olaparib, Durvalumab and Bevacizumab in Advanced FIGO Stage IV High Grade Serous Ovarian Cancer
Brief Title: NEoadjuvant Olaparib Combination OvArian Cancer Targeted Study
Acronym: NEOCATS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: AstraZeneca (Industry); Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OZM-136
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer Stage IV
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; Bevacizumab; Biosimilar Pharmaceuticals; durvalumab

STUDY DESIGN:
Intervention Model Description: Single arm, open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olaparib-Durvalumab-Bevacizumab (Experimental): Olaparib 300mg PO BID continuous dosing, Durvalumab 1500mg IV Day 1, Bevacizumab 10mg/kg IV Day 1 and 15 of a 28-day cycle Patients that respond to the therapy following 2 cycles will receive a 1 further cycle with the C3 Day 15 Bevacizumab omitted.
  Interventions: Drug: Olaparib; Drug: Bevacizumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Olaparib — Olaparib 300mg orally twice daily on a continuous dosing schedule for a maximum of 3 x 28-day cycles.
Drug: Bevacizumab — Bevacizumab 10mg/kg intravenously on Day 1 and 15 of the 28 day cycle for a maximum of 3 cycles (Cycle 3, Day 15 will be omitted).
  Other Names: biosimilar
Drug: Durvalumab — Durvalumab 1500mg intravenously on Day 1 of the 28 day cycle for a maximum of 3 cycles.

SUMMARY:
The goal of this phase 2 clinical trial is to learn if the three treatments olaparib, durvalumab and bevacizumab can treat participants with a diagnosis of stage 4 high grade serous ovarian cancer that is too advanced to undergo upfront surgery.

The main questions it aims to answer are:

Is the treatment able to shrink the cancer sufficiently for participants to undergo surgery? Is the combination of treatments safe in this neoadjuvant (before surgery) setting? This is a single arm study with no comparator arm.

Participants will receive the treatment up to 3 cycles with each drug given as follows in a 28-day cycle:

Olaparib orally on a twice daily continuous dosing schedule Durvalumab given intravenously on day 1 Bevacizumab given intravenously on day 1 and 15 (Day 15 omitted in C3)

Participants will be assessed throughout the study for safety and efficacy endpoints

DETAILED DESCRIPTION:
This is a single arm, proof of concept phase 2 study. Subjects with a suspected or confirmed diagnosis of high grade serous ovarian cancer who are not thought to be candidates for primary debulking surgery and are considered candidates for neoadjuvant chemotherapy and are not known to have BRCA mutation associated HGSOC will be considered for the trial.

Patients will be given the following triplet therapy for 2 cycles: Olaparib 300mg PO BID continuous dosing, Durvalumab 1500mg IV day 1, Bevacizumab 10mg/kg IV on day 1 and 15 of a 28-day cycle.

Patients that respond to the therapy following 2 cycles will receive 1 further cycle followed by interval cytoreductive surgery planned 3-4 weeks after completion of cycle 3 and at least 28 days from the last dose of Bevacizumab.

Following surgery, patients will revert back to standard of care (SOC) treatment and receive up to 6 cycles of chemotherapy followed by SOC recommended maintenance treatments as determined by the local treating oncology teams.

All subsequent treatments received and their response will be recorded as part of the study data collection up to and including first documented progression.

Patients that do not respond to the therapy after 2 cycles will discontinue the triplet therapy and switch to salvage standard of care treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
2. Histologically proven high grade serous ovarian/ fallopian tube or primary peritoneal cancer.
3. Chemotherapy naïve for high grade serous ovarian/ fallopian tube or primary peritoneal cancer.
4. FIGO Stage IVA/B disease not suitable for primary debulking surgery but must have the intention of proceeding to interval surgical debulking if treatment response is demonstrated
5. Patients must have disease amenable to pre-operative screening biopsies for additional translational endpoints or availability of sufficient archival tissue for additional translational endpoints including HRR pathway testing.
6. At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (or magnetic resonance imaging [MRI] where CT is contraindicated) and is suitable for repeated assessment as per RECIST 1.1. The baseline scan must be obtained within 28 days prior to the first dose of study treatment.
7. Age ≥18 years.
8. Body weight >30 kg
9. ECOG performance status 0-1 within 7 days of study registration.
10. Life expectancy of > 4 months.
11. Normal organ and bone marrow function within 14 days prior to first dose, including:

    1. Platelets ≥100x109/L
    2. Hemoglobin ≥10 g/dL with no blood transfusion in the past 28 days
    3. ANC ≥ 1.5 X 109/L
    4. Total bilirubin ≤1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome
    5. AST (SGOT) & ALT (SGPT) ≤2.5×ULN, unless liver metastases are present, in which case they must be ≤5×ULN
    6. Estimated creatinine clearance ≥51 mL/min using the Cockroft-Gault equation or based on a 24 hour urine test
12. Females of childbearing potential who are sexually active with a non-sterilized male partner must agree to use at least 1 acceptable method of contraception from the time of signing of the informed consent, throughout the period of taking study treatment and for at least 6 months after last dose of olaparib, for at least 6 months after last dose of Bevacizumab, and at least 90 days from the last dose of durvalumab, or they must totally/truly abstain from any form of sexual intercourse during these time periods.

    Non-sterilized male partners of a female patient must use male condom plus spermicide throughout this period.

    Cessation of birth control after this point should be discussed with a responsible physician. Not engaging in sexual activity for the total duration of the drug treatment and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control.
13. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1. Postmenopausal is defined as:

    1. Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    2. Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
    3. radiation-induced oophorectomy with last menses >1 year ago
    4. chemotherapy-induced menopause with >1 year interval since last menses
    5. surgical sterilisation (bilateral oophorectomy or hysterectomy)
14. Ability to understand and the willingness to sign a written informed consent document.
15. Subject's willingness and ability to comply with scheduled visits, treatment plans, on study biopsies, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Known germline BRCA1/2 mutation carriers or known somatic BRCA1/2 mutation associated HGSOC (prior to screening)
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the Triplet Combination (olaparib, durvalumab, bevacizumab).
3. Use of any other anti-cancer therapy including systemic, targeted, immunotherapy, hormonal, biological, chemotherapy, other novel agents or investigational agents within 4 weeks of registration.
4. Participation in another clinical trial with an investigational product within 4 weeks of registration
5. Previous treatment with an immune checkpoint inhibitor, including durvalumab study regardless of treatment arm assignment
6. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
7. Previously received a PARP/VEGF/PD/L-1/CTLA4 targeted therapy for this cancer diagnosis or any other cancer diagnosis in the last 5 years.
8. Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4:

   1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
   2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
   3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
   4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
9. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal breast carcinoma in situ, Stage 1, grade 1 endometrial carcinoma, or other solid tumors (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
10. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
11. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
12. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >470 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
13. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
14. Any unresolved toxicity (NCI CTCAE grade ≥2) from previous anticancer therapy, with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

    1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the sponsor.
    2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the sponsor.
15. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
16. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
17. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
18. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
19. History of leptomeningeal carcinomatosis
20. Patients with a contraindication to the use of Bevacizumab including perceived risk of perforation and uncontrolled bleeding or clotting disorder, patients with current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 28 days before study enrollment.
21. Concomitant use of known strong cytochrome P450 (CYP) 3A (CYP3A) inhibitors (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks. Concomitant use of known strong (eg, phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg, bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital land 3 weeks for other agents. Please refer to Table 3 for full details
22. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
23. History of active primary immunodeficiency. Human immunodeficiency virus (HIV) positive (positive HIV 1/2 antibodies) patients must have undetectable virology. Active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice) is not allowed.
24. Patients with known active hepatitis (i.e., hepatitis B or C). Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
25. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
26. Receipt of live attenuated vaccine within 30 days prior to enrolment
27. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g. following Hashimoto syndrome) and stable on hormone replacement therapy
    3. Any chronic skin condition that does not require systemic treatment
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study sponsor
    5. Patients with celiac disease controlled by diet alone
28. Current or prior use of immunosuppressive medication within 14 days before the first dose of enrolment. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
29. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
30. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of the triplet combination Olaparib-Durvalumab-Bevacizumab in the neoadjuvant setting in subjects with FIGO Stage IV high grade serous ovarian cancer. | Approximately 3 years, including 1 year of recruitment, 6 months treatment period, and 1 year of follow-up
  Objective Response Rate (complete response (CR) + partial response (PR)) at 8 weeks based on RECIST 1.1. as assessed by the Investigator.

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be presented as part of the final study results in a peer reviewed publication and study reports
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following final publication. No end date.